CLINICAL TRIAL: NCT02546011
Title: The Monica External Fetal Heart Rate Monitor Compared to the Standard Fetal Heart Rate Monitor
Brief Title: The Monica Fetal Heart Monitor
Status: Completed | Type: Observational
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, fruhman@slu.edu, PI, St. Louis University
Other Study IDs: 24511
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Last update posted 2016-08-05 (Estimated); Status verified 2016-08

CONDITIONS: Fetal Heart Tracing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Fetal Heart Rate Monitor — Standard of care, not part of research

SUMMARY:
The goal of this study is to compare the amount of time that the fetal heart tones are traced in babies just at or beyond viability using a traditional device compared to the Monica device.

DETAILED DESCRIPTION:
If a patient is admitted to the antepartum service and is between 24 - 28 weeks gestation, the investigators will approach the patient and inform her about the study. If the patient agrees to the study then the baby's heart tracings and contraction pattern will start to be monitored using the traditional device. If the patient would be receiving continuous fetal heart rate monitoring, then after at least 2 hours of monitoring with the traditional device, the traditional device would be replaced with the Monica device for 2 hours. After the Monica device is used for 2 hours, then the traditional device would be used once again. The entire length of the patient's participation in the study should be nor more than 6 hours.

The data collection sheet shows all data elements to be collected from the medical record. In addition it is standard of care that the monitoring strips become part of the medical records and these will also be reviewed as per the data collection sheet. Time it should take to review a patients medical record will be about 1 hour.

Total time of patient's involvement will be 7 hours.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients between 24 and 28 weeks admitted to the antepartum service

Exclusion Criteria:

* Patients with a non viable pregnancy
* Patients with multiple gestation
* Clinically Unstable patients
* Non English speaking patients

Ages: 13 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The potential participants will be on the antepartum service so we will be providing them with antepartum and obstetrical care clinically.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
To compare the amount of time that the fetal heart tones are traced in babies just at or beyond viability using a traditional device compared to the Monica device | How long can hetal heart tracings be capture continuously
  This study is to compare the amount of time that the fetal heart tones are traced in babies just at or beyond viability using a traditional device compared to the Monica device.

CONTACTS AND LOCATIONS:
Overall Officials: Gary Fruhman, MD, Principal Investigator — St. Louis University
Locations (1):
- St. Mary's Health Center, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No